CLINICAL TRIAL: NCT00110773
Title: A Randomized, Double-Blind, Placebo Controlled, Parallel Study Evaluating the Efficacy of S-Caine™ Peel (Lidocaine 7% and Tetracaine 7% Cream) to Provide Local Dermal Anesthesia for Pulsed Dye Laser Therapy in Adults
Brief Title: S-Caine™ Peel (Skin Numbing Cream) to Treat Pain During Pulsed Dye Laser (PDL) Therapy in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ZARS Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCP-42-05
Record Dates: First submitted 2005-05-12; First posted 2005-05-13 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- S-Caine Peel (Experimental)
  Interventions: Drug: S-Caine™ Peel (lidocaine and tetracaine topical cream 7%/7%)
- Placebo Peel (Placebo Comparator)
  Interventions: Drug: Placebo Peel

INTERVENTIONS:
Drug: S-Caine™ Peel (lidocaine and tetracaine topical cream 7%/7%) — S-Caine Peel, composed of a 1:1 (w:w) eutectic mixture of 7% lidocaine and 7% tetracaine, applied topically. S-Caine Peel applied at approximately 1 mm in thickness and remained on the treatment area for 20 minutes (±2 minutes).
  Other Names: Pliaglis
  Arms: S-Caine Peel
Drug: Placebo Peel — Placebo Peel applied topically at approximately 1 mm in thickness and remained on the treatment area for 20 minutes (±2 minutes).
  Other Names: Placebo
  Arms: Placebo Peel

SUMMARY:
Pulsed dye laser (PDL) on the face is painful. For this reason, local anesthesia is commonly used to eliminate or minimize the pain. S-Caine™ Peel (lidocaine 7% and tetracaine 7% cream) is a eutectic formulation of lidocaine and tetracaine. The purpose of this study is to evaluate the efficacy of S-Caine Peel for induction of local dermal anesthesia for PDL therapy in adults.

DETAILED DESCRIPTION:
This was a multi-center (5 centers), double-blind, placebo-controlled, parallel study that included 80 adults who met all the eligibility criteria and who were undergoing PDL therapy for the treatment of vascular lesions on the face.

During the screening visit, the study, including potential risks and benefits, was clearly explained to each patient, and written informed consent was obtained from each patient. The screening visit also included: evaluating eligibility criteria, obtaining a medical history (including skin type, demographic data, and concomitant medications), a brief physical examination, and a urine pregnancy test (for women of childbearing potential). The screening visit could be completed on the same day as the procedure visit.

At the procedure visit, eligible patients were assigned the next available sequential patient number. By having a patient number assigned to them, patients were randomized to receive S-Caine Peel or placebo on the facial treatment area.

The surface area of the intended treatment area was determined (up to 200 cm2). A thin layer (approximately 1 mm or the thickness of a dime) of the study drug was applied evenly across the area to be treated. The study drug was applied for 20 minutes (±2 minutes).

Immediately following removal of the study drug, the investigator performed an evaluation of skin reactions, assessing the treatment area for erythema, edema and blanching or any other adverse skin reaction.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older
* Patient elects to undergo PDL therapy for the treatment of vascular lesions on the face

Exclusion Criteria:

* Patient is pregnant or breastfeeding
* Patient has participated in a clinical trial of an unapproved drug within the previous 30 days
* Patient has participated in any clinical trial involving S-Caine Peel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-06; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 20 minutes
  Patient's evaluation of procedural pain intensity using the 100 mm Visual Analog Scale (VAS).

SECONDARY OUTCOMES:
Number of participants with adverse events | 20 minutes
  To monitor the nature and frequency of adverse events (AEs) associated with the application of S-Caine Peel

CONTACTS AND LOCATIONS:
Overall Officials: Tina Alster, MD, Principal Investigator — Washington Institute of Dermatologic Laser Surgery
Locations (3):
- United States (3):
  - Washington Institute of Dermatologic Laser Surgery, Washington D.C., District of Columbia
  - Midwest Cutaneous Research, Clinton Township, Michigan
  - Laser and Skin Surgery Center of New York, New York, New York